CLINICAL TRIAL: NCT06182540
Title: Bioavailability and Bioactivity of Mango (Poly)Phenols on Gut Health.
Brief Title: Bioavailability and Bioactivity of Mango Polyphenols.
Acronym: MANGUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Andalusian Institute of Agricultural and Fisheries Research and Training (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC/19/0097
Record Dates: First submitted 2023-11-03; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-11

CONDITIONS: Nutrition, Healthy
Keywords: Mango; Polyphenols; Ileostomy; GI tract

STUDY DESIGN:
Intervention Model Description: Acute intervention in populations with and without colon
Masking Description: Blinded analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ileostomy cohort (Experimental)
  Interventions: Dietary Supplement: Mango puree
- Non-Ileostomy cohort (Experimental)
  Interventions: Dietary Supplement: Mango puree

INTERVENTIONS:
Dietary Supplement: Mango puree — Mango puree 300g

SUMMARY:
To date however, the majority of information on bioaccessibility and bioavailability of mango phytochemicals has been generated in vitro and animal models using isolated compounds or extracts from mango leaf and mango seed kernels, which do not represent the delivery/absorption of phytochemicals from a complex food matrix such as mango puree. Consequently, a paucity of data exists on the bioavailability and metabolism of (poly)phenolic compounds following ingestion of fresh mango puree either using targeted or untargeted metabolomics approaches. Mango puree (poly)phenolic bioavailability in humans (both healthy and ilesotomists) will be investigated using both targeted and untargeted metabolomics; further we will establish the bioactivity of mango (poly)phenols with respect to gastrointestinal health. A comprehensive understanding of the bioavailability of fresh mango puree (polyp)henols, will have direct relevance to the development of any mango-based novel food products.

Acute bioavailability feeding study in two groups Ileostomists (n= 10) and health adults (N=10), as described below. Prior to attending the visit participants were asked to follow a restriction diet for 48 hours before the study and also during the 24 hours of the study clinic visit, which involved the intake of food containing low levels of polyphenols.

Ileostomists (n=10) Twenty four hours before clinic visit, the participant started a urine collection, and were asked to fast from 9pm the night before the visit (i.e. no food taken overnight and no breakfast). On the morning of the study day, the participants were asked to attend the clinic, bringing their overnight stoma bag. The 24 hr urine sample was provided, and the overnight stoma bag was removed and replaced with a new stoma bag by the participant, and passed to the researcher. A cannula was fitted in the participants arm by a qualified phlebotomist and a blood sample (~14 ml, 6 ml draw off + 8ml sample) collected. The participant was given ~300 g of mango purée to consume. Blood samples (~14 ml, 6 ml draw off + 8ml sample) were collected at hourly intervals for 8 hrs from the cannula (0, 0.5,1,1.5,2,3,4,6,8 and 24 hrs). Urine was collected between 0-4 hrs, 4-8hrs and 8-24 hrs, a fresh sample bottle was provided at each time point. Ileal samples were collected at 0-4 hrs, 4-8hrs and 8-24 hrs, the stoma bag was removed and replaced with a new stoma bag by the participant at each sampling point. A restriction diet lunch was provided to the participant after the 4 hr blood draw. After the 8 hr sample the participant was free to return home. The next morning the participant returned to the clinic and the 24 hr samples (blood, urine, ileal) collected. The urine & ileal samples were collected, and normal a normal phlebotomy draw will be used to collect the 24 hr blood sample. The participant is then finished the study was free to return to their normal diet.

Ileostomist participants each provided 4 ileal fluid samples, 4 urine samples and 10 blood samples over the sampling period.

Healthy participants (n=10) Twenty four hours before clinic visit, the participant started a urine collection, they were asked to fast from 9pm the night before the visit (i.e. no food taken overnight and no breakfast). On the morning of the study day, the participant was asked to attend the clinic. The 24 hr urine sample was collected and a faecal sample was provided. A cannula was fitted in the participants arm by a qualified phlebotomist and a blood sample (~14 ml, 6 ml draw off + 8ml sample) collected. The participant was then given ~300 g of mango purée to consume. Blood samples (~14 ml, 6 ml draw off + 8ml sample) were collected at hourly intervals for 8 hrs from the cannula (0, 0.5,1,1.5,2,3,4,6,8 and 24 hrs). Urine samples were collected between 0-4 hrs, 4-8hrs and 8-24 hrs, a fresh sample bottle was provided at each time point. A restriction diet lunch was provided to the participant after the 4 hr blood draw. After the 8 hr sample the participant was free to return home. The next morning the participant returned to the clinic and the 24 hr samples (blood, urine, faecal) collected. The urine and faecal samples were collected, and normal a normal phlebotomy draw was used to collect the 24 hr blood sample. The participant then finished the study and was free to return to their normal diet.

Healthy adult participants each provided in total 2 faecal samples, 4 urine samples and 10 blood samples over the sampling period.

ELIGIBILITY:
Inclusion Criteria (Ileostomates):

* Free-living, adult with an ileostomy, ≥1.5-years post-operative
* Aged 18-70 years at recruitment
* Non-smokers

Exclusion Criteria (Ileostomates): :

* Non-free-living adults
* Adults <18 or >70 years at recruitment
* Current smokers
* Pregnant/lactating females
* Ileostomy <1.5-year post-operative

Inclusion Criteria (Healthy adults):

* Free-living, apparently healthy adults
* Aged 18-70 years at recruitment
* Non-smokers
* No ileostomy

Exclusion criteria (Healthy adults):

* Non-free-living adults
* Adults <18 or >70 years at recruitment
* Current smokers
* Pregnant/lactating females
* Absence of gastro intestinal disease (e.g. coeliac disease; cancer)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Quantification of circulating (blood) (poly)phenols and microbially derived metabolities in participants with colon compared to without colon (ileostomates). | Change over 24 hours compared
  Quantification of polyphenols via LC-MS/MS
Quantification of urinary (poly)phenols and microbially derived metabolities in participants with colon compared to without colon (ileostomates). | Change over 24 hours
  Quantification of polyphenols via LC-MS/MS
Quantification of faecal (poly)phenols and microbially derived metabolities in participants with colon compared to without colon (ileostomates). | Change over 24 hours
  Quantification of polyphenols via LC-MS/MS

SECONDARY OUTCOMES:
Ileal fluid polyphenolic metabolites | Change over 24 hours
  Mass spectrometry analysis of In vitro gut model colonic fermentation of ileal fluid (µmol/L)
Ileal fluid microbial mediated metabolites | Change over 24 hours
  Mass spectrometry analysis of In vitro gut model colonic fermentation of ileal fluid (µmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster Univeristy, Coleraine, N.Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caceres-Jimenez S, Molinero N, Cueva C, Dobani S, Pourshahidi KL, Gill CIR, Tuohy KM, Moreno-Rojas JM, Crozier A, Bartolome B, Moreno-Arribas MV, Pereira-Caro G. Fecal fermentation of human ileal fluid after mango intake impacts on colonic microbiota and microbial (poly)phenol catabolism. Food Res Int. 2025 Dec;221(Pt 1):117217. doi: 10.1016/j.foodres.2025.117217. Epub 2025 Aug 11. PMID 41606941
- [Derived] Caceres-Jimenez S, Pereira-Caro G, Dobani S, Pourshahidi K, Gill CIR, Moreno-Rojas JM, Almutairi TM, Clifford MN, Crozier A. Interpretation of plasma pharmacokinetics and urinary excretion of phenolic metabolites and catabolites derived from (poly)phenols following ingestion of mango by ileostomists and subjects with a full gastrointestinal tract: complications associated with endogenous and ingested phenylalanine and tyrosine. Food Funct. 2025 Sep 29;16(19):7761-7778. doi: 10.1039/d5fo02745d. PMID 40928077
- [Derived] Caceres-Jimenez S, Pereira-Caro G, Dobani S, Pourshahidi K, Gill CIR, Moreno-Rojas JM, Ordonez-Diaz JL, Almutairi TM, Clifford MN, Crozier A. Bioavailability of mango (poly)phenols: An evaluation of the impact of the colon, and phenylalanine and tyrosine on the production of phenolic catabolites. Free Radic Biol Med. 2024 Nov 20;225:605-616. doi: 10.1016/j.freeradbiomed.2024.10.289. Epub 2024 Oct 18. PMID 39426756